CLINICAL TRIAL: NCT00376415
Title: A Randomized, Double-blind Placebo-controlled Phase 1 Trial of Lessertia Frutescens in Adults.
Brief Title: A Safety Study of Lessertia Frutescens in Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of the Western Cape (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R21AT001944 (NIH); R21AT001944 (NIH); TICIPS-001 (Other Grant/Funding Number: NCCIH); NCT00200772 (obsolete NCT alias)
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Drug Safety
Keywords: Lessertia frutescens; Sutherlandia frutescens; Phase 1 clinical trial; Human safety study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lessertia Fructescens (Experimental): Participants received 400mg lessertia fructescens leaf powder capsules twice daily for 3 months.
  Interventions: Drug: Lessertia Fructescens
- Placebo (Placebo Comparator): Participants received an identical placebo capsule twice daily for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lessertia Fructescens — Participants received 400mg lessertia fructescens leaf powder capsules twice daily for 3 months.
  Other Names: Sutherlandia Phytotherapy
  Arms: Lessertia Fructescens
Drug: Placebo — Participants received an identical placebo capsule twice daily for 3 months.
  Arms: Placebo

SUMMARY:
Lessertia frutescens (L.) Goldblatt & J.C. Manning (syn. Sutherlandia frutescens (L.) R. Br.), infusions and decoctions are widely used in South Africa as indigenous medicines, to combat cancer, infections and symptoms associated with AIDS. The aim of this study was to evaluate the safety of this phytotherapy in healthy adults.

DETAILED DESCRIPTION:
Objectives: Lessertia frutescens (L.) Goldblatt & J.C. Manning (syn. Sutherlandia frutescens (L.) R. Br.), infusions and decoctions are widely used in South Africa as indigenous medicines, to combat cancer, infections and symptoms associated with AIDS. The aim of this study was to evaluate the safety of this phytotherapy in healthy adults.

Design: A randomised, double blind, placebo-controlled trial to evaluate the safety of Lessertia frutescens in healthy adults.

Setting: Karl Bremer Hospital, Bellville, South Africa.

Participants: 25 adults, aged 18 to 45 years, who provided informed consent. They had no significant diseases or clinically abnormal laboratory blood profiles during screening. They had no history of allergic conditions and were not on regular medical treatment.

Intervention: 12 healthy participants were randomized to a treatment arm where they received 400mg L. frutescens leaf powder capsules twice daily (800mg/day), available as a product called Sutherlandia. 13 healthy participants were randomized to the control arm, where they received an identical placebo capsule. The trial lasted 3 months.

Outcome Measures: The primary endpoint was frequency of adverse events and the secondary endpoint, changes in physical, vital, blood and biomarker indices.

Results: There were no significant differences in general adverse events, cardiovascular, CNS, GIT, infection, allergy, malaise, most physical, haematological, biochemical or physiological parameters, between the treatment and the placebo groups (P>0.05). However, subjects consuming L. frutescens mostly reported improved appetite compared to those in the placebo group (P<0.01). Although the treatment group exhibited a lower respiration rate (P<0.04), higher platelet count (P<0.03), MCH (P<0.01), MCHC (P<0.02), total protein (P<0.03) and albumin levels (P<0.03), than the placebo group, these differences remained within the normal physiological range, and were not clinically relevant. The L. frutescens biomarker, Canavanine, was undetectable in subject plasma.

Conclusion: Overall, consumption of 800mg/day L. frutescens leaf powder capsules, was well tolerated by healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Healthy males and females between 18 and 45 years of age will:

* be informed of the nature of the study and will give written informed consent;
* have body weights within 25% of the appropriate range;
* have no significant decreases or clinically abnormal laboratory values during screening;
* have 12 lead ECG without significant abnormalities;
* be on no regular medical treatment;
* be able to communicate effectively with study personnel.

Exclusion Criteria:

* Any disease or condition which might compromise the haematopoietic, renal, endocrine, pulmonary, central nervous system, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* History of allergic conditions - asthma, urticaria and eczema.
* History of autoimmune disorders - Lupus erythematosis.
* History or presence of dyspepsia, gastric ulcer or duodenal ulcer.
* History of psychiatric disorders.
* Intake of any medication within 14 days before the start of the study.
* Recent history of alcoholism (<2 years) or consumption of alcohol within 48 hours of receiving study medication.
* Smokers who smoke more than 10 cigarettes per day and cannot refrain from smoking during the study period.
* Presence of clinically significant abnormal laboratory results during screening.
* Pregnancy or not using appropriate means of contraception.
* Use of any recreational drugs or a history of drug addiction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2004-09; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Through end of study

SECONDARY OUTCOMES:
Change in study drug biomarker levels | Through end of study
  Biomarker, Canavanine, was measured
Change in appetite | Through end of study
Change in respiration rate | Through end of study
Change in complete blood count | Through end of study
Change in serum protein levels | Through end of study
Change in serum albumin levels | Through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Haylene Nell, MBChB, Principal Investigator — Tiger Trial Centre, Karl Bremmer Hospital, Tygerberg, South Africa; Quinton Johnson, PhD, Study Director — South African Herbal Science and Medicine Institute, University of the Western Cape, Bellville, South Africa
Locations (1):
- Tiger Trial Centre, Tygerberg, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided